CLINICAL TRIAL: NCT01366690
Title: The PeerCARE Study (Peer Community-based Assistant in REtention): Effect of Peer Health Workers on People Living With HIV Not on Antiretroviral Therapy-A Randomized Trial
Brief Title: The PeerCARE Study (Peer Community-based Assistant in REtention)
Acronym: PeerCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Rakai Health Sciences Program (Other)
Responsible Party: Principal Investigator, Larry William Chang, Assistant Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00040431
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: HIV
Keywords: HIV; community health workers; randomized trial; task shifting; Uganda; retention; operations research; implementation research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Support (Experimental): Peer supporter assigned to participant.
  Interventions: Behavioral: Peer Support
- Standard of Care (No Intervention): No peer assigned. Current standard of care.

INTERVENTIONS:
Behavioral: Peer Support — A trained peer supporter is assigned to support newly HIV-positive diagnosed persons.
  Arms: Peer Support

SUMMARY:
The provision of HIV care and prevention services in resource-limited settings (RLS) entails substantial challenges due to a human resource crisis.[1] One strategy to address this human resource crisis is task shifting-the redistribution of tasks from higher trained providers to health workers with less training. Peer supporters, a group of community health workers who are people living with HIV (PLHIV), are an underutilized cadre to whom tasks can be shifted. Peers have been used extensively and effectively in HIV/AIDS programs in RLS, typically as peer educators who provide HIV prevention and education services.[2] Peers may be a potential source for not only providing care, but also impacting patient behaviors through peer counseling, education, and psychosocial support.

With the scale up of HIV counseling and testing in RLS, increasing numbers of PLHIV know their serostatus and could potentially be engaged in care and prevention services. While antiretroviral therapy (ART) is a critical component of care which has been a source of much attention, PLHIV who are not yet on ART can also benefit from being engaged in care and utilizing other evidence-based health interventions besides ART. Also, many HIV/AIDS care programs have difficulty both retaining PLHIV in care prior to ART and initiating ART in a timely fashion. Additionally, many PLHIV not yet on ART still engage in risky sexual behaviors and do not fully utilize a proven basic preventive care package (BCP) set of interventions (cotrimoxazole prophylaxis, bed nets, and safe water systems). Peers may be able to impact PLHIV not yet on ART by improving linkages to care, facilitating timely initiation of preventive interventions and ART, and decreasing risky sexual behaviors. However, well-designed and evaluated operations research is needed to assess peer support effects on these care and behavioral outcomes.

The objective of this study is to assess the impact of a peer support home visit intervention on patient engagement in care, utilization of a basic care package (BCP) of preventive care interventions, and risky sexual behaviors among people living with HIV (PLHIV) not on antiretroviral therapy (ART) through an individually randomized, operations research, community-based trial. We will compare outcomes between PLHIV who receive the peer-led intervention to those who do not. The primary outcomes will be engagement in care, BCP adherence, and condom use. The study hypotheses are as follows: (1) PLHIV who receive the peer intervention will have improved engagement in care compared to PLHIV not receiving the intervention; (2) PLHIV who receive the peer intervention are more likely to adhere to a BCP of interventions to prevent illness compared to PLHIV not receiving the intervention; (3) PLHIV who receive the peer intervention will have less risky sexual behaviors compared to PLHIV not receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Newly found to be HIV-infected through Rakai Health Sciences Program (RHSP) testing
* Agreed to receive HIV results
* Able to give consent for this study
* Age 18 years or greater

Exclusion Criteria: See above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Engagement in Care | 1 Year
Basic Care Package Adherence | 1 Year
  Adherence to a basic care package of preventive care interventions (bednets, water vessels, cotrimoxazole)
Condom Use | 1 Year
  Consistent, inconsistent, or never condom use.

SECONDARY OUTCOMES:
ART Use | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Larry William Chang, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Rakai Health Sciences Program, Entebee, Uganda

REFERENCES:
- [Derived] Monroe A, Nakigozi G, Ddaaki W, Bazaale JM, Gray RH, Wawer MJ, Reynolds SJ, Kennedy CE, Chang LW. Qualitative insights into implementation, processes, and outcomes of a randomized trial on peer support and HIV care engagement in Rakai, Uganda. BMC Infect Dis. 2017 Jan 10;17(1):54. doi: 10.1186/s12879-016-2156-0. PMID 28068935